CLINICAL TRIAL: NCT05105997
Title: Dexamethasone as a Bupivacaine Adjuvant in Ultrasound-guided Erector Spinae Plane Block for Patients Undergoing Laparoscopic Cholecystectomy: a Randomized Double-blind Study
Brief Title: Dexamethasone/ Erector Spinae Plane Block Analgesia in Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, Assistant professor of Anesthesia and Intensive Care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SM 10 2021
Record Dates: First submitted 2021-10-23; First posted 2021-11-03 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone/ Erector Spinae Plane Block (Active Comparator): Patients will receive bilateral Ultrasound-guided Erector Spinae Plane Block with bupivacaine and dexamethasone 15 minutes before skin incision.
  Interventions: Drug: Dexamethasone/ Erector Spinae Plane Block
- Erector Spinae Plane Block (Placebo Comparator): Patients will receive bilateral Ultrasound-guided Erector Spinae Plane Block with bupivacaine and one ml of normal saline 15 minutes before skin incision.
  Interventions: Drug: Erector Spinae Plane Block

INTERVENTIONS:
Drug: Dexamethasone/ Erector Spinae Plane Block — Patients will receive bilateral Ultrasound-guided Erector Spinae Plane Block with bupivacaine and dexamethasone 15 minutes before skin incision
  Arms: Dexamethasone/ Erector Spinae Plane Block
Drug: Erector Spinae Plane Block — Patients will receive bilateral Ultrasound-guided Erector Spinae Plane Block with bupivacaine and one ml of normal saline 15 minutes before skin incision.
  Arms: Erector Spinae Plane Block

SUMMARY:
Although considered a minimally invasive procedure, laparoscopic cholecystectomy (LC) frequently results in moderate to severe immediate postoperative pain.

DETAILED DESCRIPTION:
Although considered a minimally invasive procedure, laparoscopic cholecystectomy (LC) frequently results in moderate to severe immediate postoperative pain. In addition to predominant visceral pain, nearly half of all patients suffer from shoulder pain in the early postoperative period. The most likely reason is sub-diaphragmatic irritation, which is transmitted by the phrenic nerve, causing referred pain in the C4 dermatome. Due to multiple sources of pain, multimodal analgesia approaches have been used in the perioperative period following LC.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective LC under general anesthesia, ASA status I-II, aged from 18 to 65 years old of both sex

Exclusion Criteria:

* Contraindications to regional block (coagulopathy, infection at the needle insertion site, or diaphragmatic paralysis)
* Altered conscious level
* Pregnancy
* Body mass index (BMI > 35)
* Advanced hepatic or renal failure
* Chronic opioid consumption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
The intensity of postoperative pain | 24 hours after surgery
  Assessed by the verbal analog pain scale graded from 0 to 10 (0 = no pain, and 10 = the worst possible pain)